CLINICAL TRIAL: NCT06279975
Title: Investigative Neurological Study With Pupillometric Evaluation os a Clinical Tool in Patients Declared Brain Dead (INSPECT) - a Prospective Quality Control Study
Brief Title: Pupillometric Evaluation in Patients Declared Brain Dead - a Prospective Quality Control Study
Acronym: INSPECT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2023-01275; am23Sutter2
Record Dates: First submitted 2023-11-22; First posted 2024-02-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Brain Death; Adults
Keywords: Pupillometry; Brain Death; Diagnosis
MeSH Terms: conditions — Brain Death; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: non-invasive device-supported, automated pupillometry — non-invasive device-supported, automated pupillometry with a precise quantitative measurement of the pupils within the range of micrometers

SUMMARY:
The aim of the study is to verify the reliability of the current purely clinical examination of the pupils (without the support of a pupillometer) in the context of clinically suspected brain death, compared to the results of a non-invasive, automated, and highly precise monocular pupillometric examination.

DETAILED DESCRIPTION:
This prospective quality control study will evaluate the reliability of the clinical exam regarding pupils' reaction to light (as performed by two board certified physicians in Neurology and/or Intensive Care Medicine) as recommended by the SAMW guidelines for brain death diagnosis (SAMW-guidelines) when compared to the results of a noninvasive automated and highly-precise pupillometry in adult patients with clinically suspected brain death. Automated pupillometric measurements will be performed by the PI (RS), or the co-investigator (Dr. Pascale Grzonka) using the NeurOptics® NPi®-200 pupillometer system immediately before and after the standardized diagnostic workup for suspected brain death. In addition, demographics, clinical characteristics , treatment and laboratory data from the patients examined will be anonymously collected.

ELIGIBILITY:
Inclusion Criteria:

* Suspected diagnosis of brain death
* Brain death diagnostic procedures planned
* Treated at the intensive care unit at the University Hospital Basel (USB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population is defined as all adult patients (i.e. ≥18 years of age) treated on the intensive care unit at the University Hospital Basel (USB) in whom the treating physicians suspect brain death and plan to perform brain death diagnostic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Reliability of clinical examination of pupils in patients with suspected brain death | baseline (2 hours before start of brain death evaluation) and 5 hours (2 hours after end of brain death evaluation)
  Determination of the reliability of the current purely clinical examination of the pupils (without the support of a pupillometer) in the context of clinically suspected brain death compared to the results of a noninvasive, automated, and highly precise pupillometric examination (measurement of the discordance between automated analyses of pupillary light reflex by a hand-held pupillometer and visual examination without pupillometer support in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Intensive care unit at the University Hospital Basel, Basel, Canton of Basel-City
  - University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: No